CLINICAL TRIAL: NCT01640457
Title: A Prospective Randomized Multicentre Phase I/II Clinical Trial to Evaluate Safety and Efficacy of NOVOCART® Disc Plus Autologous Disc Chondrocyte Transplantation (ADCT) in the Treatment of Nucleotomized and Degenerative Lumbar Discs to Avoid Secondary Disease
Brief Title: Safety and Efficacy With NOVOCART® Disc Plus (ADCT) for the Treatment of Degenerative Disc Disease in Lumbar Spine
Acronym: NDisc
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tetec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-1102
Record Dates: First submitted 2012-05-16; First posted 2012-07-13 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Intervertebral Disc Displacement; Intervertebral Disc Degeneration
Keywords: degenerative disc; herniated disc; sequestrectomy; Autologous Disc Chondrocyte Transplantation; nucleotomy; safety; efficacy; treatment; lumbar spine; low back pain; adjacent degenerative disc; black disc; NOVOCART
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NDplus (Experimental): NOVOCART® Disc plus (Autologous Disc Chondrocyte Transplantation System)
  Interventions: Drug: NOVOCART® Disc plus
- NDbasic (Placebo Comparator): NOVOCART® Disc basic (media with no active cell component)
  Interventions: Device: NOVOCART® Disc basic
- Sequestrectomy only (SC) (No Intervention): Sequestrectomy (standard of care)

INTERVENTIONS:
Drug: NOVOCART® Disc plus — Autologous Disc Chondrocyte Transplantation System (ADCT)
  Arms: NDplus
Device: NOVOCART® Disc basic — ADCT (Media with no active cell component)
  Arms: NDbasic

SUMMARY:
NOVOCART® Disc plus is being investigated to explore its clinical applicability, safety and efficacy in the repair of a herniated disc with an indication for an elective sequestrectomy, and of the adjacent degenerated disc, if present. The objective of this clinical study is to provide basis for a confirmatory study design (endpoints, methodologies) (Phase II), and to develop a safety profile (Phase I). This study further aims at developing and validating known and new biologic markers for the quality and clinical efficacy of the product as requested in the context of identity, purity and potency characteristics of the medicinal/investigational product.

DETAILED DESCRIPTION:
This is a classical Phase II study with an implicated Phase I part. The Phase I/II combination study is a non-confirmatory study aimed at gathering preliminary clinical information on NOVOCART® Disc plus used in a new indication in the repair of a herniated disc. It will be conducted in a prospective, multicenter, unmasked, clinical trial including 120 subjects randomized to NOVOCART® Disc plus (NDplus, 60 subjects), media NOVOCART® Disc basic with no active cell component (NDbasic, 36 subjects) and to standard of care (SC) sequestrectomy as control (24 subjects). 24 patients will be enrolled in Phase I of the study (12 NDplus, 12 NDbasic) and 96 patients in Phase II (48 NDplus, 24 NDbasic, 24 SC).

All subjects will be evaluated at 1.5-, 3-, 6-, 12-, 24-, 36-, 48-months post-t0 examination in the SC study arm and 1.5-, 3-, 6-, 12-, 24-, 36-, 48-months post-t5 examination in the NDplus and NDbasic study arms, and then 5 years post-t0/t5 to collect long-term clinical data. Efficacy measurements for functional improvement will be evaluated among NDplus, NDbasic and SC. Physiological effects observed from MRI measurements will be compared between appropriate treatments depending on expected treatment mechanisms. Safety data of NDplus will be combined with NDbasic to contrast against SC on procedure related risks and NDplus against NDbasic and SC together on graft-related adverse experiences.

To optimize the usefulness of clinical information, data collected in the study may be analyzed and reviewed continuously. Early findings may be used to modify the study design when deemed appropriate and acceptable by the Sponsor's medical advisors. Data-driven adaptive actions include but are not limited to stopping enrollment early. The Sponsor will inform regulatory bodies, Ethic Committees, and investigators before implementing study design modifications.

Cells and tissues collected from this study will be used in other in vitro-controlled experiments aimed at developing and validating known and novel biologic markers to quantify cell quality in the context of identity, purity and potency. Prognostic values of these biologic markers will be examined by correlating them with clinical data collected in this study.

The study will follow each subject for a total of five years post-t0 examination in the SC study arm and post-t5 examination in the NDplus and NDbasic study arms to obtain long-term performance data.

Patients must have a single-level acute disc herniation with an indication for an elective sequestrectomy. They may further have corresponding disc degeneration in the proximal adjacent segment (Pfirrmann Score Stage 3-4). A total of 120 adults will be enrolled in this study.

Each patient will remain in the study for 5 years post t0/t5 examination to complete the planned follow-up phase. It is expected to take 6 years and five months to collect all required data for this study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a disc herniation with back and/or leg pain (radicular pain)
2. The patient has an indication for sequestrectomy according to the guidelines of DGNC and DGOOC
3. The patient is between 18-60 years of age.
4. The patient is physically and mentally able to participate in the study, and is able to understand the study, its goals and the possible risk factors involved. The patient is willing and able to participate in the follow-up visit plan at the study site and is able to understand and to complete study-relevant questionnaires in German language.
5. The patient is sufficiently informed about this trial orally and in writing. S/he had enough time for consideration, is willing to participate in the study and gives her/his written in-formed consent.
6. The patient confirms that s/he did not participate in a clinical study 90 days prior study inclusion. S/he agrees to refrain from participating in another clinical study during the NOVOCART® Disc Study and for another 90 days after study termination

Radiological Inclusion Criteria

Patients must meet all of the following criteria to be considered for enrollment in the NOVO-CART® Disc study.

1. The patient has a single-level lumbar disc herniation
2. The patient has more than 50% remaining disc height in the herniated disc in comparison to unaffected discs in the lumbar spine. If all discs show degenerative signs, disc height has to be at least 5 mm
3. The patient has no obvious signs of osteophytes and no end plate sclerosis in the lumbar segment to be treated with NOVOCART® Disc plus oder NOVOCART® Disc basic

Patients without adjacent degenerative disc (HD):

4. The adjacent proximal disc has no degenerative signs according to Pfirrmann Score stage 3 to 5.

Patients with adjacent degenerative disc (AAD):

4. The patients has additional degenerative signs in the proximal adjacent lumbar level ac-cording to Pfirrmann 3-4, but no more than 25% disc height reduction

Exclusion Criteria:

1. The patient has had a previous surgery at the lumbar level(s) and has been treated with NOVOCART® Disc plus oder NOVOCART® Disc basic.
2. The patient had a past recurrent disc herniation treated with sequestrectomy of the relevant disc.
3. The patient has any degenerative muscular or neurological condition that would interfere with evaluation of outcome measures including but not limited to Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis, muscular dystrophy and myelopathic diseases of different causes.
4. BMI > 35 kg/m2
5. The patient has current or recent history of illicit drug, nicotine (more than 20 cigarettes per day) or alcohol abuse or dependence
6. CRP > 10mg/dl
7. The patient is pregnant, breastfeeding or actual planning to become pregnant. Female patients must be either at least two years postmenopausal or using one of the following means of birth control during the treatment phase, i.e. to transplantation

   * surgical sterility
   * double barrier methods, e.g. condom or diaphragm in combination with spermicide
   * intrauterine contraceptive device
   * bilateral vasectomy of sexual partner at least 90 days prior to enrolment in combination with barrier methods (e.g. condom or diaphragm)
   * birth control pill
8. The patient has a history of known allergies or a suspicion of allergies to any of the NO-VOCART® Disc plus oder basic product components including hyaluronan, polyethylenglycol or albumin
9. Immune defects or the affinity for infections of known or unknown causes
10. The patient has a active systemic or local microbial infection, eczematization or inflammable skin alterations at the site of surgery (including Protozoonosis: Babesiosis, Trypanosomiasis (e.g. Chagas-Disease), Leishmaniasis, persistent bacterial infections, like Brucellosis, spotted and typhus fever, other Rickettsiosis, Leprosy, Recurrent Fever, Melioidosis or Tularaemia).
11. The patient is unable to undergo magnetic resonance imaging (MRI)
12. The patient has a history or a suspicion of a disease with chronically inflammable character, as rheumatoid arthritis, gout, pseudo-gout, metabolic bone diseases, Crohn's disease, ulcerative colitis, lupus erythematosus, or other autoimmune disorders
13. Known osteoporosis
14. The patient has a primary hyperparathyroidism or hyperthyroidism, has chronic renal failure or has had previous fragility fractures.
15. Systemic connective tissue or collagen disease
16. Hereditary ocular degenerations with unclear diagnosis, retinopathies based on connective tissue-defined causes, macular corneal dystrophy, (based on the fact that the human cornea expresses cartilage specific proteins as essential functional elements and thus may serve as an indicator for paralleling degenerative events in various cartilaginous tissues)
17. The patient has immune suppression
18. The patient has a history of blood coagulation disease of different genesis, including known haemorrhagic diathesis of unknown cause
19. The patient had undergone chemo or radiotherapy within the past 5 years, or had any cancer other than non-melanoma skin cancer treated with curative intent within the past 5 years
20. Known diabetes, drug treated
21. Ulterior concomitant diseases or functional impairments of specific organs, which exclude study participation by the assessment of the investigator
22. The patient is a prisoner

Radiological Exclusion Criteria

• 1. The patient has apparent degenerative changes in the lumbar spine as determined by Modic Changes 2-3 2. The patient has one or more dysplastic vertebral bodies within the lumbar spine 3. The patient has a sacralised lumbar vertebra LWK5 at the level to be treated with NOVOCART® Disc plus oder NOVOCART® Disc basic 4. The patient has previous or acute spondylodiscitis 5. Segmental instability (spondylolisthesis > 5 mm) or translation > 3 mm 6. The patient has a isthmic spondylolisthesis, ankylosing spondylitis or spondylolysis 7. The patient has lumbar scoliosis (> 11° deformation). 8. The patient has previous trauma, discography or any other surgical intervention at the lumbar spine .

9. The patient has previous compression or burst fracture at the level(s) to be treated with NOVOCART® Disc plus or NOVOCART® Disc basic 10. The patient has a central spinal canal stenosis with evidence of a narrowing of < 8 mm (by MRI, sagittal ) 11. The patient has a spinal tumor 12. The patient has metabolic bone disease 13. The patient has facet ankylosis or severe facet degeneration. 14. The patient has a lumbar kyphosis

Intra-surgery (tissue explant/sequestrectomy) Exclusion Criteria

1. Extensive damage of the Anulus, which subsequently poses a significantly greater risk of recurrence.

Exclusion criteria determined after tissue explant/sequestrectomy

1. HIV infection
2. Treponema pallidum (syphilis) infection
3. active hepatitis B or C infection

Exclusion Criteria prior Transplantation/Implantation

1. Recurrent disc herniation after surgery and prior transplantation/implantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2018-11-01 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) to 12-months follow-up
  Primary efficacy variable.
  Early evaluation for efficacy will be performed when all patients completed scheduled 12-months follow-up visit (Interim analysis).
Oswestry Disability Index (ODI) | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) to 24-months follow-up
  Primary efficacy variable.
  Primary evaluation for efficacy will be performed when all patients completed scheduled at 24-months follow-up visit (Interim analysis).
Oswestry Disability Index (ODI) | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) to 60-months follow-up
  Primary efficacy variable.
  Final analysis will be performed when all patients completed scheduled 60-months follow-up visit.

SECONDARY OUTCOMES:
MRI-signal (disc height, disc volumetry, signal intensity) | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Oswestry Disability Index | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
VAS for back pain and leg pain | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Health-related quality of life as measured by the SF-36 | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Healthy Questionnaire EQ-5D | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Neurological status | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Functional status | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Return to work (days) | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Analgesic Medication Use during the previous 14-day-time period | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 60-months follow-up
  Secondary efficacy variable
  Early evaluation for efficacy will be performed at 12-months follow-up, primary evaluation for efficacy will be performed at 24-months follow-up, and final analysis will be performed at 60-months follow-up.
Physician assessments of ease of transplantation | transplantation
  Outcome to quantify feasibility of procedure
  When all NDplus and NDbasic patients completed transplantation procedure.
Surgical parameters, including length of procedure | Sequestrectomy and transplantation
  Outcome to quantify feasibility of procedure
  When all enrolled patients completed sequestrectomy and if applicable transplantation procedure.
Prevalence of subsequent surgical interventions | 12-months post-operation
  Outcome to Quantify Safety
  A subsequent surgical intervention is defined as any invasive procedure performed at the index level to treat the same condition (herniation) or other conditions resulted from the transplantation/implantation procedure within the 12-month period post-operation.
Any unanticipated adverse event | Baseline assessment 1<45d pre-sequestrectomy up to 60-months follow-up at any scheduled and unscheduled visit
  Outcome to Quantify Safety
Specific laboratory parameters according to product compatibility and availability: CRP, IL-6, LTE4 | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 1,5-months follow-up
  Outcome to Quantify Safety (Phase I only)
  At sequestrectomy, 2h-, 6h-, 24h-, 36h- post surgery, transplantation, direct after transplantation, 6h-, 12h-, 18h-, 24h-, 30h-, 36h-, 42h-, 48h- post transplantation, 3 and 6 weeks post transplantation
Histology of the tissue explant | Sequestrectomy
  Outcome to Develop and Validate Biological Markers
Gene expression by quantitative realtime PCR of expanded cells, and cell culture medium metabolites during expansion | Transplantation
  Outcome to Develop and Validate Biological Markers
Biomarkers of blood and urine samples (SOX9, MMP-3, collagen type I, collagen type II, collagen type X, IL-1, aggrecan, BMP receptor Ia, BSP-2, FLT-1, collagen crosslinks, and yet to be defined additional elements) | Baseline assessment 1<45d pre-sequestrectomy, pre-transplantation (90 +/- 15d post-sequestrectomy) up to 24-months follow-up
  Outcome to Develop and Validate Biological Markers

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joerg Meisel, Professor, Principal Investigator — Hospital "BG-Kliniken Bergmannstrost, Halle"; Claudius Thomé, Professor, Principal Investigator — University Hospital for Neurosurgery Innsbruck
Locations (10):
- University Hospital for Neurosurgery Innsbruck, Innsbruck, Tyrol, Austria
- Germany (9):
  - Charité Universitätsmedizin, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - University Hospital Duesseldorf, Düsseldorf
  - Universitätsmedizin, Göttingen
  - Hospital "BG-Kliniken Bergmannstrost", Halle
  - SHG Klinikum, Idar-Oberstein
  - Städtisches Klinikum, Karlsruhe
  - Berufsgenossenschaftliche Unfallklinik, Murnau am Staffelsee
  - St. Franziskus Hospital, Münster

REFERENCES:
- [Derived] Tschugg A, Michnacs F, Strowitzki M, Meisel HJ, Thome C. A prospective multicenter phase I/II clinical trial to evaluate safety and efficacy of NOVOCART Disc plus autologous disc chondrocyte transplantation in the treatment of nucleotomized and degenerative lumbar disc to avoid secondary disease: study protocol for a randomized controlled trial. Trials. 2016 Feb 26;17(1):108. doi: 10.1186/s13063-016-1239-y. PMID 26920137